CLINICAL TRIAL: NCT01786083
Title: Depression and Anxiety Symptoms Reduction and Perceived Wellbeing Improvement in Female Primary Caregivers of Chronically Ill Patients by the Application of Problem Solving Technique by Primary Health Care Nurses
Brief Title: Caring for Family Caregivers:a Research-action Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Preventive Services and Health Promotion Research Network (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 070489
Record Dates: First submitted 2013-02-01; First posted 2013-02-07 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Depressive Symptoms; Anxiety; Emotions
Keywords: family caregivers; dependency; Problem Solving Technique; home based nursing
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Experimental): Application of Problem Solving Technique
  Interventions: Behavioral: Application of Problem Solving Technique
- No counseling (No Intervention): Usual care by caregiver

INTERVENTIONS:
Behavioral: Application of Problem Solving Technique
  Arms: Lifestyle counseling

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the Problem Solving Technique (PST) in reducing symptoms of anxiety and depression among primary caregivers of chronically ill patients.

And also to describe and evaluate the process carried out by nurses when implementing the PST as a useful tool for care for family caregivers.

DETAILED DESCRIPTION:
Background: In Spain, home care for the chronically ill and their family caregivers should be a priority in health and social policies due to the aging of the population and the progressive increase in dependent individuals. In our case, 88% of healthcare within dependency care is provided by the family and only 12% by health professionals. The family requires comprehensive and multidisciplinary ongoing care, in which the primary healthcare nurse plays a leading role. One of the areas involved is home-based nursing and counselling for family caregivers, in order to improve the quality of the care provided and to prevent issues arising that may adversely affect the caregiver's life.

Method: This is a research-action study with a mixed analysis methodology. Quantitative analysis was used to evaluate the effectiveness of the Problem Solving Technique in reducing symptoms of anxiety and depression among family caregivers. The clinical trial involved a control and experimental group and pre-post intervention measurements, using the Goldberg scale of anxiety and depression. The sample consisted of 122 caregivers who presented one of these positive subscales. The technique's application process was evaluated for the qualitative analysis, with a content analysis of the records of 10 nurses performing the experimental intervention.

ELIGIBILITY:
Inclusion Criteria:

Caregivers of chronically ill patients included in the ATDOM programme, who at the time of the intervention had a positive score on the Goldberg scale for anxiety and/or depression.

Exclusion Criteria:

Professional caregivers

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-09; Primary Completion 2009-09 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Anxiety | Two years
  Goldberg Scale
Depression | Two years
  Goldberg scale
perceived wellbeing levels | two years
  Primary caregiver's Emotional health(NOC 2506)

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Health Centers, Tarragona Province, Tarragona, Tarragona, Spain

REFERENCES:
- See also: Social and Family Wellbeing Department of the Catalan Government — http://www20.gencat.cat/portal/site/bsf/menuitem.7fca6ecb84d307b43f6c8910b0c0e1a0/?vgnextoid=fdb6859e616a4210VgnVCM1000008d0c1e0aRCRD&vgnextchannel=fdb6859e616a4210VgnVCM1000008d0c1e0aRCRD